CLINICAL TRIAL: NCT06855732
Title: Pain Self-Management Intervention to Reduce Pain & Improve MOUD Engagement in Primary Care: A Randomized Trial
Brief Title: Pain Self-Management and Treatment Engagement for Patients Taking Opioids
Acronym: TREETOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin Winstanley, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24080167; RM1DA055311 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain; Opioid Use Disorder; Opioid Misuse and Addiction
Keywords: pain; opioid; primary care; behavioral health
MeSH Terms: conditions — Chronic Pain; Opioid-Related Disorders; Behavior, Addictive; Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to either PSM or Usual Care.
  The intervention will be completed in 12 weeks and will take place between the baseline and 3-month (post-intervention) visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (Active Comparator): Usual care refers to the standard of care that patients receive at their primary care clinic.
  Interventions: Behavioral: Usual Care
- Pain Self-Management (PSM) (Experimental): PSM is a manualized pain self-management behavioral intervention tailored to patients with chronic pain and opioid misuse/OUD. PSM consists of 10 intervention sessions delivered via phone or web-based communication platform. Sessions will be led by a staff interventionist.
  Interventions: Behavioral: Pain Self-Management

INTERVENTIONS:
Behavioral: Usual Care — Usual care refers to the standard of care that patients receive at their primary care clinic.
  The standard of care for patients is to discuss chronic pain with their providers at their discretion, and for providers to offer buprenorphine for OUD and/or provide referrals to specialty addiction treatment programs in the local community.
  Participants will continue to have access to usual care for chronic pain, which could include pain clinic visits, physical therapy, medication (e.g., gabapentin), and/or seeing a counselor, psychiatrist, or psychologist.
  The study protocol will not interfere with usual clinical care.
  Arms: Usual Care
Behavioral: Pain Self-Management — PSM is a manualized behavioral intervention tailored to patients in primary care with opioid misuse/OUD. The PSM intervention that consists of ten sessions/modules.
  Participants will be offered a total of 10 PSM sessions, delivered weekly over a 12-week intervention period starting from the date of study enrollment.
  A trained staff interventionist will lead the 60-minute sessions using a participant study manual that outlines the content for all 10 sessions.
  The first two sessions, "Introduction" and "Navigating Conversations About Opioids", are mandatory. Participants can choose the order of the remaining 8 sessions, prioritizing those they are most interested in. Additional session topics are: Stress Management and Your Pain, Relaxation Techniques to Help Your Pain, Thinking Differently About Your Pain, Sleeping Better to Help Your Pain, Physical Activity and Your Pain, Mood and Your Pain, and Communicating with Others.
  Arms: Pain Self-Management (PSM)

SUMMARY:
The goal of this study is to learn if Pain Self-Management (PSM) can improve chronic pain care in individuals with opioid misuse or opioid use disorder (OUD) The main questions it aims to answer are:

* Does PSM help participants manage their chronic pain more effectively?
* Does PSM help participants engage in treatment for opioid use?

Researchers will compare PSM to standard care to see if PSM is effective in managing chronic pain and engagement in treatment.

Participants will:

* Take part in the PSM program or receive standard care for 12 weeks after enrolling in the study
* Complete surveys every 3 months for 9 months (total of 4 visits)

Participants will receive compensation for participating in the study.

There are risks associated with participating in the study, including breach of confidentiality and psychological distress caused by discussing difficult topics.

DETAILED DESCRIPTION:
This is randomized trial of a pain self-management (PSM) intervention for chronic pain tailored to individuals with opioid misuse or opioid use disorder (OUD) as compared to usual care. The investigators hypothesize that PSM will be effective in improving both reducing pain and improving MOUD engagement among individuals with co-occurring opioid misuse/OUD and chronic pain.

This is a multisite trial recruiting from primary care clinics located in Pennsylvania, West Virginia and Maryland.

Interventions: Participants will be randomized to either PSM or Usual Care.

Pain Self-Management (PSM): PSM is a manualized pain self-management behavioral intervention tailored to patients with chronic pain and opioid misuse/OUD. PSM consists of 10 intervention sessions delivered via phone or web-based communication platform. Sessions will be led by a staff interventionist.

Usual Care (UC): Usual care or "treatment as usual" refers to the standard of care that patient participants receive at their primary care clinic. The standard of care for patients is to discuss issues related to chronic pain and opioid use with their providers and to receive clinical care for these conditions.

Study Duration: ~27 months (18 months of recruitment + 9 months follow-up) Participant Duration: 9 months

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Adults at least 18 years old
2. Ability to speak, read, and understand English
3. Capable of providing informed consent
4. Access to phone and/or internet
5. Current (defined as at least 1 primary care visit in the past 3 years) or new (confirmed appointment) primary care patient at a participating clinic
6. Must meet criteria for OUD or opioid misuse based on at least one of the following:

   1. OUD Misuse Screening score of 3 or more (sometimes or more) on at least one of the questions
   2. Meets criteria for DSM-5 Opioid Use Disorder on MINI-J
   3. Documented diagnosis of Opioid use Disorder (OUD)
7. Have bothersome (Grade 2) or high impact chronic pain (Grade 3), based on the Graded Chronic Pain Scale-Revised (GCPS-R)

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Under 18 years of age
2. Have cancer-related pain
3. Are currently in jail, prison, overnight/residential facility as required by court of law or have pending legal action that could prevent participation in study activities
4. Have received prescribed, administered, or dispensed MOUD (buprenorphine, methadone, naltrexone) as maintenance treatment for OUD (excluding acute or short-term (< 7 days) use of these medications to manage opioid withdrawal or pain management) within the past 90 days
5. Had an intentional suicide attempt within the past 3 months

The investigators will not exclude individuals with common comorbidities, such as depression, anxiety, or alcohol, methamphetamine, and other substance use disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Interference as Assessed by the PROMIS SF v1.0 - Pain Interference 4a at 3 months Post-baseline | Baseline, 3 Months
  The PROMIS Pain Interference - Short Form 4a is a validated, self-report 4-item tool assessing pain interference over the past 7 days. The PROMIS SF v1.0 - Pain Interference 4a consists of 4 questions and uses a 5-point scale, ranging from 1 (not at all) to 5 (very much). The total raw score equals the sum the values of the response to each question. The raw score is converted to a T-score. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like pain interference, a T-score of 60 is one SD worse than average. That is, a person has more problems with pain hindering activities. By comparison, a pain interference T-score of 40 is one SD better than average.
  Change = 3 month score - baseline score

SECONDARY OUTCOMES:
Change from Baseline in Overall Pain as Assessed by the PEG at 3 months Post-baseline | Baseline, 3 Months
  The Pain, Enjoyment, and General Activity (PEG) Scale is a validated, self-report 3-item tool assessing pain intensity and interference over the past week. The PEG scale consists of 3 separate numerical scales. Each scale has ratings ranging from 0-10. The PEG score is calculated by averaging the three numbers; a higher score indicates greater pain.
  Change = 3 month score - baseline score
Change from Baseline in Pain Catastrophizing as Assessed by the Pain Catastrophizing Questionnaire-6-item at 3 months Post-baseline | Baseline, 3 Months
  The Pain Catastrophizing Scale is a validated, self-report 6-item tool assessing assess pain catastrophizing for chronic pain. The PCS-6 uses a 5-point scale, ranging from 0 (not at all) to 4 (all the time). The total score ranges from 0 to 24, with higher score representing greater catastrophic thinking.
  Change = 3 month score - baseline score
Proportion of Participants that Engage in MOUD Treatment at 3 months Post-baseline | Baseline, 3 Months
  Proportion of individuals who self-reported having filled a prescription for or were administered or dispensed any MOUD (methadone, buprenorphine, naltrexone)
Number of Days Participants took MOUD at 6-months Post-baseline | 6 Months
  MOUD: methadone, buprenorphine, naltrexone.
  Measured by self-report and medical chart extraction.
Change from Baseline in Self-Efficacy at 3 months Post-baseline | Baseline, 3 Months
  Change in self-efficacy for managing symptoms as measured by the Pain Self-Efficacy Questionnaire (PSEQ).
  The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire developed to assess the confidence people with ongoing pain have in performing activities while in pain. The PSEQ is applicable to all persisting pain presentation. It enquires into the level of self-efficacy regarding a range of functions, including household chores, socializing, work, as well as coping with pain without medication.
  A raw score is presented with a range from 0 - 60, where high scores indicate greater levels of confidence in dealing with pain. High scores are strongly associated with clinically-significant functional levels and provide a useful gauge for evaluating outcomes in chronic pain patients.
  Change = 3 month score - baseline score
Number of Days Non-prescribed Opioids were Used in the past 30 days as Assessed by the Modified ASI at 3-months Post-baseline | 3 Months
  The modified ASI is a validated, self-report tool which includes questions from the Addiction Severity Index section on drug and alcohol use and includes questions about specific opioids used. The number of days in the last 30 that a participant reports using heroin, fentanyl, and/or opioid analgesics (percocet, oxycodone, oxycontin, vicodin, dilaudid, hydrocodone, hydromorphone, morphine, or codeine) will be summed for the outcome "Number of days non-prescribed opioids were used in the past 30 days." Number of days may range from 0 to 90.
Total score on the IMPOWR Opioid Misuse Screening scale at 3 months Post-baseline | 3 Months
  The IMPOWR Opioid Misuse Screening scale is an exploratory, self-report scale consisting of 4 questions about the use of prescribed pain medications. Each question response ranges from Never (0) to Almost Always (4) with a possible summed score ranging from 0 to 16, with higher scores indicating more severe misuse.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Winstanley, PhD, Principal Investigator — University of Pittsburgh
Locations (16):
- United States (16):
  - Renaissance Family Practice - Hampton Office, Allison Park, Pennsylvania
  - Renaissance Family Practice - RIDC Office, Blawnox, Pennsylvania
  - Renaissance Family Practice - Glenshaw Office, Glenshaw, Pennsylvania
  - Renaissance Family Practice - Millvale Office, Pittsburgh, Pennsylvania
  - Community Medicine, Inc., Pittsburgh, Pennsylvania
  - UPMC General Internal Medicine-Montefiore, Pittsburgh, Pennsylvania
  - Renaissance Family Practice - Aspinwall Office, Pittsburgh, Pennsylvania
  - UPMC General Internal Medicine-Shadyside (Shea Medical Center), Pittsburgh, Pennsylvania
  - Renaissance Family Practice - Harmarville Office, Pittsburgh, Pennsylvania
  - UPMC General Internal Medicine-Turtle Creek, Turtle Creek, Pennsylvania
  - Renaissance Family Practice - Penn Hills Office, Verona, Pennsylvania
  - UPMC General Internal Medicine-South, West Mifflin, Pennsylvania
  - St. Joseph's Rural Health Clinic (WVU Medicine), Buckhannon, West Virginia
  - Harpers Ferry Family Medicine (WVU Medicine), Harpers Ferry, West Virginia
  - WVU Medicine University Town Centre, Morgantown, West Virginia
  - WVU Medicine Primary Care, Shepherdstown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the HEAL Public Access and Data Sharing Policy (https://www.nih.gov/research-training/medical-research-initiatives/heal-initiative/research/heal-public-access-data-sharing-policy) and data for this study will be available to the public through the IMPOWR Dissemination Education and Coordination Center (IDEA-CC) (https://heal.nih.gov/research/clinical-research/integrative-management-chronic-pain).
Supporting Information: Study Protocol, SAP
Time Frame: De-identified data will be made available within 18 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Access to trial IPD may be made available to individuals that submit a request along with the required documents to the IMPOWR data committee. Data access requires approval by the IMPOWR data committee and the individual must agree to comply with the data sharing policies of IMPOWR and HEAL.
URL: https://heal.nih.gov/research/clinical-research/integrative-management-chronic-pain